CLINICAL TRIAL: NCT05468970
Title: Single-center Real World Prospective Observational Study of Clinical Features, Treatment Patterns, and Survival of Bone and Soft Tissue Tumors
Brief Title: Study on Clinical Features, Treatment Mode and Survival of Bone and Soft Tissue Tumors
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, Associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-12
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Bone and Soft Tissue Tumors; Clinical Features
MeSH Terms: conditions — Soft Tissue Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO Intervention — NO Intervention

SUMMARY:
It is planned to prospectively collect, collate and report real-world clinical data of BSTS patients treated in our hospital in the next ten years to evaluate the changes in clinical characteristics, treatment patterns and survival information of these patients, in order to provide reference for clinical treatment and research of this type of tumor.

DETAILED DESCRIPTION:
It is planned to prospectively collect, collate and report real-world clinical data of BSTS patients treated in our hospital in the next ten years to evaluate the changes in clinical characteristics, treatment patterns and survival information of these patients, in order to provide reference for clinical treatment and research of this type of tumor. This study is a single-center, prospective, real-world observational study that plans to enroll all eligible patients. Basic information, treatment methods, and prognostic information of these patients were collected.

ELIGIBILITY:
Inclusion Criteria:

All ages, male and female.

The pathological diagnosis of BSTS in our hospital was a subtype.

Has received at least one hospitalization in this hospital.

The target lesions could be evaluated according to the efficacy evaluation criteria of solid tumor (RECIST; Version 1.1) Measure diameter changes.

Exclusion Criteria:

No definite pathology.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bone and soft tissue tumors receiving inpatient treatment in Henan Tumor Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to approximately 120months
  Pathologically confirmed events leading to death
6/5000 Progression-free survival | Up to approximately 48months
  The time from the first use of the treatment to the observation of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided